CLINICAL TRIAL: NCT01340404
Title: A Multicenter Study Comparing the Results of Allogeneic Stem Cell Genoidentical in Children With Sickle Cell Anemia and Cerebral Vascular Disease Detected by Transcranial Doppler
Brief Title: Allogeneic Genoidentical Stem Cell Transplantation in Children With Sickle-cell Anemia and Cerebral Vasculopathy
Acronym: DREPAGREFFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P071247
Record Dates: First submitted 2011-04-21; First posted 2011-04-22 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-11

CONDITIONS: Sickle Cell Anemia; Cerebrovascular Accident
MeSH Terms: conditions — Anemia, Sickle Cell; Stroke | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem Cell Transplantation (Experimental)
  Interventions: Procedure: Stem cell transplantation
- Transfusion program (Active Comparator)
  Interventions: Procedure: Transfusion program

INTERVENTIONS:
Procedure: Stem cell transplantation — Stem cell transplantation
  Arms: Stem Cell Transplantation
Procedure: Transfusion program — Transfusion program
  Arms: Transfusion program

SUMMARY:
The aim of this study is to demonstrate that cerebral velocities assessed by transcranial doppler (TCD) are more significantly decreased by SCT than by long-term transfusion program A multicenter, national, non-randomized, prospective study of paired cohort will be conducted, with 2 groups of exposed (SCT) and non-exposed (TP) patients.

DETAILED DESCRIPTION:
The aim of this study is to demonstrate that cerebral velocities assessed by transcranial doppler (TCD)are more significantly decreased by SCT than by long-term transfusion program A multicenter, national, non-randomized, prospective study of paired cohort will be conducted, with 2 groups of exposed (SCT) and non-exposed (TP) patients. Sixty-three patients will be enrolled, namely 21 sickle-cell patients in the "SCT" group and 42 in the "Transfusion Program (TP)" group

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell anemia patients (SS/Sb0)
* < 15 years old
* History of abnormal transcranial doppler (TCD) (≥ 200 cm/sec)
* Siblings from the same parental couple
* Parents amenable to Human Leucocyte Antigen (HLA) typing, SCT if an HLA-identical sibling is available or to long-term transfusion program

Exclusion Criteria:

* Sickle cell patients older than 15 years
* no history of abnormal transcranial doppler (TCD) (≥ 200 cm/sec)
* no sibling from the same parental couple
* parents averse to HLA typing, SCT if an HLA-identical sibling is available or to long-term transfusion program

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2010-12; Primary Completion 2013-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Cerebral vasculopathy | 1 year
  velocity in the artery with highest velocity

SECONDARY OUTCOMES:
ischemic lesions on magnetic resonance imaging (MRI) | 1 year
  percentage of patients with ischemic lesions on magnetic resonance imaging (MRI)
stenoses on magnetic resonance imaging (MRI) | 1 year
  percentage of patients with stenoses on magnetic resonance imaging (MRI)
normalisation of arterial velocities | 12 months
  percentage of patients at 1 year with velocities normalization on transcranial doppler (TCD)(< 170 cm/sec)

OTHER OUTCOMES:
cognitive dysfunction | 12 months
  the scale of cognitive dyfunction depends on the child's age : definition of dysfunction uses the WISC-4, WPPSI-4 or WAIS-3 according to age

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Bernaudin, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- CHIC, Créteil, France

REFERENCES:
- [Derived] Bernaudin F, Verlhac S, Peffault de Latour R, Dalle JH, Brousse V, Petras E, Thuret I, Paillard C, Neven B, Galambrun C, Divialle-Doumdo L, Pondarre C, Guitton C, Missud F, Runel C, Jubert C, Elana G, Ducros-Miralles E, Drain E, Taieb O, Arnaud C, Kamdem A, Malric A, Elmaleh-Berges M, Vasile M, Leveille E, Socie G, Chevret S; DREPAGREFFE Trial Investigators. Association of Matched Sibling Donor Hematopoietic Stem Cell Transplantation With Transcranial Doppler Velocities in Children With Sickle Cell Anemia. JAMA. 2019 Jan 22;321(3):266-276. doi: 10.1001/jama.2018.20059. PMID 30667500
- [Derived] Chevret S, Verlhac S, Ducros-Miralles E, Dalle JH, de Latour RP, de Montalembert M, Benkerrou M, Pondarre C, Thuret I, Guitton C, Lesprit E, Etienne-Julan M, Elana G, Vannier JP, Lutz P, Neven B, Galambrun C, Paillard C, Runel C, Jubert C, Arnaud C, Kamdem A, Brousse V, Missud F, Petras M, Doumdo-Divialle L, Berger C, Freard F, Taieb O, Drain E, Elmaleh M, Vasile M, Khelif Y, Bernaudin M, Chadebech P, Pirenne F, Socie G, Bernaudin F. Design of the DREPAGREFFE trial: A prospective controlled multicenter study evaluating the benefit of genoidentical hematopoietic stem cell transplantation over chronic transfusion in sickle cell anemia children detected to be at risk of stroke by transcranial Doppler (NCT 01340404). Contemp Clin Trials. 2017 Nov;62:91-104. doi: 10.1016/j.cct.2017.08.008. Epub 2017 Aug 15. PMID 28821470